CLINICAL TRIAL: NCT03914274
Title: Importance of Sock Type in the Development of Foot Lesions on Low-difficulty, Short Hikes
Brief Title: Adequate Sock to Avoid Hiking Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Ana María Pérez Pico, Principal Investigator, University of Extremadura
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: AMPPico
Record Dates: First submitted 2019-03-17; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Skin Lesion
Keywords: Sport Injury; Technical socks; Temperature; Hiking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Thermometer "FTN" "Medisana", precision 0.18º C), (No Intervention): Temperatures were taken with an infrared thermometer "FTN" "Medisana", precision 0.18º C.
  The temperature will be taken into account to see if it will vary according to the socket used as the temperature is a favoring element of dermic injuries on the feet.
- Non-elastic tape measure (No Intervention): Perimeter was measured with a flexible, non-elastic tape measure "Lawton 18-0160", precision 1 mm.
  The measurement of the feet perimeters will be taken into account to see if it will vary according to the socket used and related to injuries in the feet.
- Bascule (No Intervention): Weight was measured using scales ("Tanita" UM-076, precision 0.1kg). The scale is used to control the weight of the participants in order to find out their body mass index since the weight can influence the appearance of lesions on the feet.
- Altimeter (No Intervention): Height was measured using the weight rod of different scales "SECA 704", precision 1 mm) The altimeter is used to measure the participants in order to find out their body mass index.
- Socks (Experimental): Socks were of two types: technical socks, designed for high performance sports use "Lurbel brand, models Tierra and Set", and non-technical socks for everyday use. The socks had different composition: "Tierra:50% regeneractiv, 25% cool-teak, 17% polyamide ions, 8% lycra"; "Set:75% cotton, 17% polyamide, 8% lycra" and "cotton: 98% cotton, 2% elastane".
  Different socks were given to the participants to see if the different compositions influenced the appearance of injuries in a short route route and little difficulty
  Interventions: Device: Technical sock
- Geographical Position System Garmin "ETREX" 20 (No Intervention): The height range and the pace hikers were controlled with a Garmin "ETREX" 20X Geographical Position System

INTERVENTIONS:
Device: Technical sock — Socks were of two types: technical socks, designed for high performance sports use (Lurbel brand, models Tierra and Set), and non-technical socks for everyday use. The socks had different composition: Tierra (50% regeneractiv, 25% cool-teak, 17% polyamide ions, 8% lycra); Set (75% cotton, 17% polyamide, 8% lycra) and cotton (98% cotton, 2% elastane).
  Arms: Socks

SUMMARY:
Foot lesions can be developed during hiking because of external factors. This makes it important to study the effect of hiking equipment on lesion development.

This study analyzes the extrinsic factors involved in the appearance of injuries at the feet during the realization of a route of low difficulty and short travel. 33 participants wore cotton not technicians socks in his two feet, were used like control socks and 76 participants wore technical socks "Tierra" and "Set" one on each foot.

DETAILED DESCRIPTION:
Socks it used as an indispensable element to protect the foot of injuries during sports practice. The different compositions of socks can influence the appearance of injuries. The technical socks are designed for high-performance sports use ("Lurbel" brand, models "Tierra" and "Set"), and non-technical socks (cotton) for everyday use. The socks had different composition: "Tierra" (50% regenerative, 25% cool-teak, 17% polyamide ions, 8% lycra); "Set" (75% cotton, 17% polyamide, 8% lycra) and cotton (98% cotton, 2% elastane). The technical socks had reinforced weave in the toe, metatarsal and heel areas.

ELIGIBILITY:
Inclusion Criteria:

* The admission criteria were: be of legal age, have no current health problems that would hinder or prevent participation in the hike, and carry a backpack weighing less than 3 kg. Participants were asked to use specific hiking footwear (light, flexible, soft-soled, with good grip and breathable material) (low top hiking shoes), based on earlier studies 38-40. They were also asked to do the entire hike following the instructions of an experienced guide and to not remove their footwear or socks before examination by a podiatrist.

Exclusion Criteria:

* Not meet any inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2015-10-10 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05-28 (Actual)

PRIMARY OUTCOMES:
lesions in foot developed during the hike | The development of the injuries in a single day of sport activity was observed: kilometer 0 of the route, kilometer 14.5 of the route and kilometer 29.6 of the route.
  All dermal lesions that developed during the walk (both keratopathies with keratinization disorder and dermatopathies without keratinization disorder) Blister, Injury, (Erosion & chafing), Reddened skin, Urticaria, Crevice, Heloma, all the muscle injuries that developed during the walk (Pain, Inflammation, Muscle discomfort or Sprain) and all the lesions in the skin were analyzed. the nails that developed during the walk, both traumatic and non-traumatic (onycopathies) Onychocryptosis, Subungual hematoma.

SECONDARY OUTCOMES:
Temperature | The temperature was measured in three occasions in a single day: kilometer 0 of the route, kilometer 14.5 of the route and kilometer 29.6 of the route
  Were mearusedTemperatures in different parts of foot with an infrared thermometer (FTN "Medisana", precision 0.18º C). Three measurements were done and their media was calculated.
Perimeter | The perimeter was measured in three occasions in a single day: kilometer 0 of the route, kilometer 14.5 of the route and kilometer 29.6 of the route
  Perimeter in different parts of foot with a flexible, non-elastic tape measure (Lawton 18-0160, precision 1 mm).Three measurements were done and their media was calculated. Three measurements were done and their media was calculated.
Weight | The weight was measured in three occasions in a single day: kilometer 0 of the route, kilometer 14.5 of the route and kilometer 29.6 of the route
  Weight was measured using scales (Tanita UM-076, precision 0.1kg).Three measurements were done and their media was calculated.
Height at the start of the route for calculate "BMI" | The height onli was measured at the start of the walk in a single day: kilometer 0 of the route
  Height was measured using the weight rod of differents scales (SECA 704, precision 1 mm). Three measurements were done and their media was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Mayordomo, Dr, Study Director — Universidad de Extremadura

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wannop JW, Worobets JT, Ruiz R, Stefanyshyn DJ. Footwear traction and three-dimensional kinematics of level, downhill, uphill and cross-slope walking. Gait Posture. 2014;40(1):118-22. doi: 10.1016/j.gaitpost.2014.03.004. Epub 2014 Mar 13. PMID 24684947
- [Background] Fattorini L, Pittiglio G, Federico B, Pallicca A, Bernardi M, Rodio A. Workload comparison between hiking and indoor physical activity. J Strength Cond Res. 2012 Oct;26(10):2883-9. doi: 10.1519/JSC.0b013e318242a61e. PMID 22158090
- [Background] Brandenburg WE, Locke BW. Mountain medical kits: epidemiology-based recommendations and analysis of medical supplies carried by mountain climbers in Colorado. J Travel Med. 2017 Mar 1;24(2). doi: 10.1093/jtm/taw088. PMID 28395094
- [Background] Serrano MA, Canada J, Moreno JC. Ultraviolet exposure for different outdoor sports in Valencia, Spain. Photodermatol Photoimmunol Photomed. 2011 Dec;27(6):311-7. doi: 10.1111/j.1600-0781.2011.00620.x. PMID 22092735
- [Background] Pigman J, Sullivan W, Leigh S, Hosick PA. The Effect of a Backpack Hip Strap on Energy Expenditure While Walking. Hum Factors. 2017 Dec;59(8):1214-1221. doi: 10.1177/0018720817730179. Epub 2017 Sep 11. PMID 28892419
- [Background] Anderson LS Jr, Rebholz CM, White LF, Mitchell P, Curcio EP 3rd, Feldman JA, Kahn JH. The impact of footwear and packweight on injury and illness among long-distance hikers. Wilderness Environ Med. 2009 Fall;20(3):250-6. doi: 10.1580/08-WEME-OR-196R2.1. PMID 19737037
- [Background] Dahl KD, Wang H, Popp JK, Dickin DC. Load distribution and postural changes in young adults when wearing a traditional backpack versus the BackTpack. Gait Posture. 2016 Mar;45:90-6. doi: 10.1016/j.gaitpost.2016.01.012. Epub 2016 Jan 22. PMID 26979888
- [Background] Jacobson BH, Wright T. A field test comparison of hiking stick use on heartrate and rating of perceived exertion. Percept Mot Skills. 1998 Oct;87(2):435-8. doi: 10.2466/pms.1998.87.2.435. PMID 9842582
- [Background] Brennan FH Jr, Jackson CR, Olsen C, Wilson C. Blisters on the battlefield: the prevalence of and factors associated with foot friction blisters during Operation Iraqi Freedom I. Mil Med. 2012 Feb;177(2):157-62. doi: 10.7205/milmed-d-11-00325. PMID 22360060
- [Background] Schoffl V, Morrison A, Hefti U, Ullrich S, Kupper T. The UIAA Medical Commission injury classification for mountaineering and climbing sports. Wilderness Environ Med. 2011 Mar;22(1):46-51. doi: 10.1016/j.wem.2010.11.008. Epub 2010 Nov 16. PMID 21377118
- [Background] Schoffl V, Morrison A, Schoffl I, Kupper T. The epidemiology of injury in mountaineering, rock and ice climbing. Med Sport Sci. 2012;58:17-43. doi: 10.1159/000338575. Epub 2012 Jul 18. PMID 22824837
- [Background] Kirkham S, Lam S, Nester C, Hashmi F. The effect of hydration on the risk of friction blister formation on the heel of the foot. Skin Res Technol. 2014 May;20(2):246-53. doi: 10.1111/srt.12136. Epub 2014 Mar 20. PMID 24645912
- [Background] Knapik JJ, Reynolds K, Barson J. Influence of an antiperspirant on foot blister incidence during cross-country hiking. J Am Acad Dermatol. 1998 Aug;39(2 Pt 1):202-6. doi: 10.1016/s0190-9622(98)70075-1. PMID 9704829
- [Background] Van Tiggelen D, Wickes S, Coorevits P, Dumalin M, Witvrouw E. Sock systems to prevent foot blisters and the impact on overuse injuries of the knee joint. Mil Med. 2009 Feb;174(2):183-9. doi: 10.7205/milmed-d-01-8508. PMID 19317200
- [Background] Choi SC, Min YG, Lee IS, Yoon GH, Kang BR, Jung YS, Cho JP, Kim GW. Injuries associated with the 580 km university student grand voluntary road march: focus on foot injuries. J Korean Med Sci. 2013 Dec;28(12):1814-21. doi: 10.3346/jkms.2013.28.12.1814. Epub 2013 Nov 26. PMID 24339714
- [Background] Zhong W, Xing MM, Pan N, Maibach HI. Textiles and human skin, microclimate, cutaneous reactions: an overview. Cutan Ocul Toxicol. 2006;25(1):23-39. doi: 10.1080/15569520500536600. PMID 16702052
- [Background] Arezes PM, Neves MM, Teixeira SF, Leao CP, Cunha JL. Testing thermal comfort of trekking boots: an objective and subjective evaluation. Appl Ergon. 2013 Jul;44(4):557-65. doi: 10.1016/j.apergo.2012.11.007. Epub 2013 Jan 12. PMID 23317756
- [Background] Tayel AA, El-Tras WF, Abdel-Monem OA, El-Sabbagh SM, Alsohim AS, El-Refai EM. Production of anticandidal cotton textiles treated with oak gall extract. Rev Argent Microbiol. 2013 Oct-Dec;45(4):271-6. doi: 10.1016/S0325-7541(13)70036-1. PMID 24401783
- [Background] Najafi B, Mohseni H, Grewal GS, Talal TK, Menzies RA, Armstrong DG. An Optical-Fiber-Based Smart Textile (Smart Socks) to Manage Biomechanical Risk Factors Associated With Diabetic Foot Amputation. J Diabetes Sci Technol. 2017 Jul;11(4):668-677. doi: 10.1177/1932296817709022. Epub 2017 May 17. PMID 28513212
- [Background] DiLiberto FE, Baumhauer JF, Nawoczenski DA. The prevention of diabetic foot ulceration: how biomechanical research informs clinical practice. Braz J Phys Ther. 2016 Nov 16;20(5):375-383. doi: 10.1590/bjpt-rbf.2014.0195. PMID 27849290
- [Background] Coughlin SS, Hatzigeorgiou C, Anglin J, Xie D, Besenyi GM, De Leo G, Stewart J, Wilkins T. Healthy lifestyle intervention for adult clinic patients with type 2 diabetes mellitus. Diabetes Manag (Lond). 2017;7(2):197-204. PMID 28794802
- [Background] Gonzalez-Vargas S, Cortes-Reyes E, Marino-Isaza F. [Prevalence of musculoskeletal injuries in racing skaters in Villavicencio, Colombia]. Rev Salud Publica (Bogota). 2017 May-Jun;19(3):347-354. doi: 10.15446/rsap.v19n3.62976. Spanish. PMID 30183939
- [Background] Janssen L, Allard NAE, Ten Haaf DSM, van Romburgh CPP, Eijsvogels TMH, Hopman MTE. First-Aid Treatment for Friction Blisters: "Walking Into the Right Direction?". Clin J Sport Med. 2018 Jan;28(1):37-42. doi: 10.1097/JSM.0000000000000424. PMID 28452830
- [Background] ElMakki Ahmed M, Tamimi AO, Mahadi SI, Widatalla AH, Shawer MA. Hallux ulceration in diabetic patients. J Foot Ankle Surg. 2010 Jan-Feb;49(1):2-7. doi: 10.1053/j.jfas.2009.07.005. PMID 20123279
- [Background] Jagoda A, Madden H, Hinson C. A friction blister prevention study in a population of marines. Mil Med. 1981 Jan;146(1):42-4. No abstract available. PMID 6783997
- [Background] Knapik JJ, Hamlet MP, Thompson KJ, Jones BH. Influence of boot-sock systems on frequency and severity of foot blisters. Mil Med. 1996 Oct;161(10):594-8. PMID 8918120
- [Background] Herring KM, Richie DH Jr. Friction blisters and sock fiber composition. A double-blind study. J Am Podiatr Med Assoc. 1990 Feb;80(2):63-71. doi: 10.7547/87507315-80-2-63. PMID 2304016
- [Background] Herring KM, Richie DH Jr. Comparison of cotton and acrylic socks using a generic cushion sole design for runners. J Am Podiatr Med Assoc. 1993 Sep;83(9):515-22. doi: 10.7547/87507315-83-9-515. PMID 8289142
- [Background] Worthing RM, Percy RL, Joslin JD. Prevention of Friction Blisters in Outdoor Pursuits: A Systematic Review. Wilderness Environ Med. 2017 Jun;28(2):139-149. doi: 10.1016/j.wem.2017.03.007. PMID 28602272
- [Background] Simpson KM, Munro BJ, Steele JR. Backpack load affects lower limb muscle activity patterns of female hikers during prolonged load carriage. J Electromyogr Kinesiol. 2011 Oct;21(5):782-8. doi: 10.1016/j.jelekin.2011.05.012. Epub 2011 Jun 25. PMID 21705231
- [Background] Frederick EC. Kinematically mediated effects of sport shoe design: a review. J Sports Sci. 1986 Winter;4(3):169-84. doi: 10.1080/02640418608732116. PMID 3586110
- [Background] Perez-Pico AM, Marcos-Tejedor F, Iglesias-Sanchez MJ, Acevedo RM. Importance of Footwear for Preventing Xerosis and Hyperkeratosis in Older People with Psychiatric Disorders Living in an Institution. Int J Environ Res Public Health. 2018 Mar 24;15(4):584. doi: 10.3390/ijerph15040584. PMID 29587357
- [Background] Peters P, Runge J. [Electronic plantar pressure measurements in different types of moutaineering boots]. Sportverletz Sportschaden. 2001 Jun;15(2):40-4. doi: 10.1055/s-2001-14816. German. PMID 11475620
- [Background] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Background] Boulware DR, Forgey WW, Martin WJ 2nd. Medical risks of wilderness hiking. Am J Med. 2003 Mar;114(4):288-93. doi: 10.1016/s0002-9343(02)01494-8. PMID 12681456
- [Background] Heggie TW, Heggie TM. Viewing lava safely: an epidemiology of hiker injury and illness in Hawaii Volcanoes National Park. Wilderness Environ Med. 2004 Summer;15(2):77-81. doi: 10.1580/1080-6032(2004)015[0077:vlsaeo]2.0.co;2. PMID 15228059
- [Background] Niedermeier M, Einwanger J, Hartl A, Kopp M. Affective responses in mountain hiking-A randomized crossover trial focusing on differences between indoor and outdoor activity. PLoS One. 2017 May 16;12(5):e0177719. doi: 10.1371/journal.pone.0177719. eCollection 2017. PMID 28520774
- [Background] Niedermeier M, Grafetstatter C, Hartl A, Kopp M. A Randomized Crossover Trial on Acute Stress-Related Physiological Responses to Mountain Hiking. Int J Environ Res Public Health. 2017 Aug 11;14(8):905. doi: 10.3390/ijerph14080905. PMID 28800067
- [Background] Bogerd CP, Rechsteiner I, Wust B, Rossi RM, Bruhwiler PA. The effect of two sock fabrics on physiological parameters associated with blister incidence: a laboratory study. Ann Occup Hyg. 2011 Jun;55(5):510-8. doi: 10.1093/annhyg/meq099. PMID 21669907
- [Background] McWhorter JW. The effects of loaded versus unloaded activities on foot volumetrics in older healthy adults. N Am J Sports Phys Ther. 2008 Feb;3(1):34-40. PMID 21509138
- [Background] Dirksen G, Bachmann PA. [Occurrence of rota- and coronavirus as a cause of neonatal calf diarrhea in the Federal Republic of Germany]. Berl Munch Tierarztl Wochenschr. 1977 Dec 15;90(24):475-7. No abstract available. German. PMID 202239
- [Background] Dao H Jr, Kazin RA. Gender differences in skin: a review of the literature. Gend Med. 2007 Dec;4(4):308-28. doi: 10.1016/s1550-8579(07)80061-1. PMID 18215723
- [Background] Leveque JL, Corcuff P, de Rigal J, Agache P. In vivo studies of the evolution of physical properties of the human skin with age. Int J Dermatol. 1984 Jun;23(5):322-9. doi: 10.1111/j.1365-4362.1984.tb04061.x. PMID 6746182

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT03914274/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT03914274/ICF_001.pdf